CLINICAL TRIAL: NCT04202627
Title: Biomarker Development in LGMD2i
Acronym: MLB-01-001
Status: Completed | Type: Observational
Sponsor: ML Bio Solutions, Inc. (Industry)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20018755
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Muscular Dystrophies; Limb Girdle Muscular Dystrophy
Keywords: LGMD; FKRP; Clinical Research; ML Bio Solutions; Limb Girdle Muscular Dystrophy; Limb girdle muscular dystrophy type R9 (LGMD R9); LGMD2i
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophies, Limb-Girdle; Muscular Dystrophy, Limb-Girdle, Type 2I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and Tissue samples will be taken for biomarker development and retained for future research. No clinical diagnosis will be given to patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of this natural history study is to define the key LGMD2i phenotypes as measured by standard clinical outcome assessments (COAs), and to validate a muscle biomarker for LGMD2i to support therapeutic development.

DETAILED DESCRIPTION:
Limb Girdle Muscular Dystrophy (LGMD) 2i is an autosomal recessive form of LGMD that is due to missense mutations in the Fukutin-related protein (FKRP) gene. Patients develop progressive proximal muscle weakness that leads to loss of ambulation. Patients will also commonly develop a cardiomyopathy and respiratory compromise.

There are promising new therapies that have been developed and as a result therapeutic trials are approaching.

The rationale for this study is to define appropriate COAs for LGMD2i, which will facilitate therapeutic development and ensure properly powered clinical trials. In addition, measurement of dystroglycan in muscles represents a potential muscle biomarker that could be used in early phase clinical trials as a measure of target engagement. The clinical utility of changes in dystroglycan has not been validated in human samples.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10-65 at enrollment
* Clinically affected (defined as weakness on bedside evaluation in either a limb-girdle pattern, or in a distal extremity)
* A genetically confirmed mutation in FKRP (LGMD2i)
* Willing and able to give informed consent and follow all procedures and requirements

Exclusion Criteria:

* Any other illness that would interfere with the ability to undergo safe testing or would interfere with interpretation of the results in the opinion of the site investigator.
* History of a bleeding disorder, platelet count <50,000, current use of an anticoagulant.
* Positive pregnancy test
* A 10-meter walk time of <4 seconds

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be identified through self-selection and direct recruitment options. Participants will be identified from the population of individuals who are followed at the neuromuscular clinics. Participants will also be solicited from the Global FKRP registry.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
10-Meter walk (10 MWT) -mobility | Through study completion at 12 months
  The 10 MWT will be used to determine the ambulatory Cohort for of all subjects. For the purposes of this study, the definitions for ambulation are as follows:
  * Cohort A: completes the 10 MWT unaided in ≥ 4 to ≤ 12 seconds
  * Cohort B: completes the walk unaided in > 12 seconds or is non-ambulatory
100-Meter Timed Test (100m) - mobility | Through study completion at 12 months
  The 100m timed test is designed to capture maximal ambulatory capacity. The participant will be asked to complete 4 full laps around 2 cones set 25 meters apart as quickly and as safely as possible, including running if able. This will not be assessed in participants with a 10-meter walk time greater than 12 seconds.
NSAD- Motor performance | Through study completion at 12 months
  North Star Assessment for Dysferlinopathy (NSAD) is a functional scale specifically designed to measure motor performance in individuals with LGMD. It consists of 29 items that are considered clinically relevant items from the North Star Ambulatory Assessment and the Motor Function Measure 20 with a maximum score of 54 and higher scores indicate higher functional abilities.
Timed up-and-go (TUG) - mobility | Through study completion at 12 months
  The TUG is an assessment used to evaluate functional ambulation, balance, and fall risk. The fastest time to rise from a chair, walk 3 meters, and return to sitting independently without an assistive device will be recorded. This will not be assessed in Cohort B participants.
FVC - Pulmonary function | Through study completion at 12 months
  The total amount of air exhaled during the forced expiratory volume test (Forced vital capacity - FVC) will be assessed in a sitting position only.
Timed 4 stair Climb (4SC) - mobility | Through study completion at 12 months
  The 4SC quantifies the time required for the participant to ascend 4 standard steps. This will not be assessed in participants with a 10 meter walk time greater than 12 seconds.
9 Hole Peg Test (9HPT) - distal upper extremity function | Through study completion at 12 months
  The 9HPT is a quantitative measure of distal upper extremity function. It measures the time required for patients to place 9 pegs in the 9 holes on the board and then remove them as quickly as possible.
Performance of Upper Limb (PUL 2.0) - limb function | Through study completion at 12 months
  The PUL is a tool designed for assessing upper limb function in persons with neuromuscular disorders. It was developed as a conceptual framework reflecting the progression of weakness and natural history of functional decline in Duchenne muscular dystrophy (DMD). There are 22 scored items; a score of 42 indicates the highest level of independent function and 0 the lowest.
Hand Held Dynamometry (HHD) - isometric strength | Through study completion at 12 months
  HHD using the MicroFET2 myometer will be utilized to capture isometric strength in target muscle groups. Maximum strength in kilograms will be reported for each muscle group provided a continuous scale variable for analysis.

SECONDARY OUTCOMES:
To develop clinical outcome assessments for LGMD2i | Through study completion at 12 months
  To determine the sensitivity of the COAs to longitudinal disease progression

OTHER OUTCOMES:
To validate potential biomarkers | Baseline, Month 6
  To develop a reliable measure of dystroglycosylation in human skeletal muscle by using fresh tissue biopsy.
  A muscle biopsy will be collected at baseline and 6 months from the right tibialis anterior. The biopsy site will be uniform between investigators. The investigators will utilize a 14-gauge Supercore biopsy instrument to take a total of three aspirations from the same site.
To understand the change from baseline in muscle mass using Magnetic Resonance Imaging | Baseline, Month 6, Month 12
  To understand the change from baseline in muscle mass using Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas E Johnson, MD, Principal Investigator — Virginia Commonwealth University
Locations (11):
- United States (10):
  - University of California Irvine, Irvine, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Atrium Health, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
- Copenhagen Neuromuscular Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No